CLINICAL TRIAL: NCT00656097
Title: A Randomized, Single-blind, Controlled, Monocentric Phase II Trial to Compare the Safety and Neutralizing Activity of Simulated Rabies Post-exposure Prophylaxis With CL184 in Combination With Rabies Vaccine vs. HRIG or Placebo in Combination With Rabies Vaccine in Healthy Adult Subjects
Brief Title: A Randomized Phase II Trial to Compare the Safety and Neutralizing Activity of CL184 in Combination With Rabies Vaccine vs. HRIG or Placebo in Combination With Rabies Vaccine in Healthy Adult Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Crucell Holland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RAB-M-A003
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-09

CONDITIONS: Rabies
Keywords: Rabies post-exposure prophylaxis
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): CL184 combined with rabies vaccination
  Interventions: Biological: CL184
- B (Active Comparator): HRIG combined with rabies vaccination
  Interventions: Biological: HRIG
- C (Placebo Comparator): Placebo combined with rabies vaccination
  Interventions: Biological: Placebo matching CL184

INTERVENTIONS:
Biological: CL184 — CL184 20 IU/kg intramuscularly on Day 0; in conjunction with rabies vaccine on Days 0, 3, 7, 14, and 28
  Arms: A
Biological: HRIG — HRIG 20 IU/kg intramuscularly on Day0; in conjunction with rabies vaccine on Days 0, 3, 7, 14, and 28
  Arms: B
Biological: Placebo matching CL184 — Placebo intramuscularly on Day0; in conjunction with rabies vaccine on Days 0, 3, 7, 14, and 28
  Arms: C

SUMMARY:
The aim of this study is to evaluate the safety of the monoclonal antibody cocktail CL184 in combination with rabies vaccine compared with human rabies immune globulin (HRIG) or placebo in combination with rabies vaccine in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects free of obvious health-problems or with stable condition
* Male or female subjects aged ≥19 to ≤65 years
* BMI between ≥18 and ≤30 kg/m2

Exclusion Criteria:

* Prior history of active or passive rabies immunization
* Clinically significant acute illness or infection within 2 weeks before first dosing based on the clinical judgment of the investigator
* History and/or family history of clinically significant immunodeficiency or auto-immune disease
* Any clinically significant history of known or suspected anaphylaxis or hypersensitivity reaction
* Chronic administration of immunosuppressants or other immune-modifying drugs within 6 months before the first dose of investigational medicinal product

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2008-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 42 days

SECONDARY OUTCOMES:
Rabies virus neutralizing activity | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: C. James Kissling, MD, Principal Investigator — MDS Pharma Services, 621 Rose Street, Lincoln, NE 68502, USA
Locations (1):
- MDS Pharma Services , USA, Lincoln, Nebraska, United States